CLINICAL TRIAL: NCT03821038
Title: International, Multicenter, Randomized, Double-blinded, Placebo-controlled Study of Recombinant Interleukin-7 (CYT107) to Restore Absolute Lymphocyte Counts (ALC) in Patients With Sepsis
Brief Title: Recombinant Interleukin-7 (CYT107) to Restore Absolute Lymphocyte Counts in Sepsis Patients
Acronym: IRIS-7-C&D
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PK issue detected after bolus IV route administration
Sponsor: Revimmune (Industry)
Collaborators: Washington University School of Medicine (Other); University Hospital, Limoges (Other); Emerald Clinical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRIS-7-C&D
Record Dates: First submitted 2019-01-24; First posted 2019-01-29 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Sepsis, Severe
Keywords: Sepsis; IL-7; lymphocytopenia
MeSH Terms: conditions — Sepsis; Lymphopenia | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: International, multicenter, randomized, double-blinded placebo- controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Open-label pharmacist will prepare masked syringes for the ICU
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CYT107 (Experimental): Intravenous (IV) administration of CYT107 at 10 μg/kg twice a week for 3 weeks
  Interventions: Biological: CYT107
- Placebo (Placebo Comparator): Intravenous (IV) administration of the same volume of NaCl 0.9% twice a week for 3 weeks
  Interventions: Drug: Placebos

INTERVENTIONS:
Biological: CYT107 — IV twice a week at 10µg/kg for 3 weeks
  Other Names: human recombinant glycosylated Interleukin-7
  Arms: CYT107
Drug: Placebos — IV twice a week at the same volume for 3 weeks
  Other Names: saline solution
  Arms: Placebo

SUMMARY:
This phase II randomized study will assess the effect of receiving IV recombinant human IL-7 (CYT107) versus placebo in lymphopenic sepsis patients

The aim is to confirm the immune cell reconstitution observed in other studies and other patient populations among which the IRIS-7 A&B study which was conducted in the same patient population.

DETAILED DESCRIPTION:
Lymphopenic sepsis Patients will be randomized 3:1 to receive either:

a) Intravenous (IV) administration of CYT107 at 10 μg/kg twice a week for 3 weeks or b) IV placebo (normal saline).

The effect of CYT107 on Lymphocyte and various T cell populations will be documented with a focus on the first 29 days.

Stopping rules will apply if ALC increases to >2.5 times the upper limit of normal range.

The IRIS-7C & D studies will be conducted at multiple sites in France and the United States. All sites will use the same study design and similar study protocol for a common statistical analysis of 40 evaluable participants.

ELIGIBILITY:
Inclusion Criteria:

1. A written, signed informed consent, by the patient or the patient's legally authorized representative
2. Participants with an absolute lymphocyte count (ALC) ≤ 900 cells/mm3, at two time points at least twelve hours apart, following diagnosis of vasopressor dependent sepsis and,

   1. the second time point should not be performed earlier than 48 hours after sepsis diagnosis,
   2. study drug treatment initiation is required no later than 120 hours (up to 5 days) after the last qualifying ALC ≤ 900 cells/mm3 measure, and
   3. the average value of the two qualifying ALC counts will serve as a baseline to express the percent increase at day 29, or at hospital discharge.
3. Patients in the ICU with onset of vasopressor dependent sepsis defined as hypotension requiring treatment with any vasopressor(s) for at least 6 hours to maintain a systolic pressure ≥ 90 mmHg or a mean arterial pressure ≥65 mmHg AND at least 1 of the 2 organ dysfunction criteria below:

   1. Acute respiratory failure defined as the need for invasive mechanical ventilation for at least 24 hours to support pulmonary function
   2. Acute kidney injury defined as creatinine > 2.0 mg/dL (based on new abnormal result following onset of sepsis) OR urine output < 0.5 mL/kg/hr for > 4 hours despite adequate fluid resuscitation. In the presence of pre-existing impairment of renal function (defined as a serum creatinine concentration >2 times the upper limit of the normal reference range prior to the onset of sepsis), the patient must meet the other organ dysfunction criteria.
4. Anticipated hospital duration of up to approx. three weeks after initiating study drug treatment to allow 6 study drug administrations (Days 18 or 19 would be final dose)
5. This study permits the re-enrollment of a participant who may have been discontinued as a pre-treatment screen failure and/or prior to study drug treatment.
6. Age and reproductive status:

   1. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment
   2. Women must not be breastfeeding
   3. Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of treatment with CYT107 plus 5 half-lives of CYT107 (the terminal half-life of CYT107 is up to 2 days) plus 30 days (duration of ovulatory cycle) for a total of 2 months post-treatment completion.
   4. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with CYT107 plus 5 half-lives of CYT107 plus 90 days (duration of sperm turnover) for a total of 7 months post-treatment completion. In addition, male participants must be willing to refrain from sperm donation during this time.
   5. Azoospermic males are exempt from contraceptive requirements.
   6. WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements but still must undergo pregnancy testing.

Exclusion Criteria:

1. Cancer with current chemotherapy or radiotherapy (receipt of chemotherapy or radiotherapy for cancer within the last 6 weeks). All patients with current, or history of, hematologic malignancy (including, but not limited to, ALL, AML, CLL, CML, etc.) or lymphoma will be excluded, regardless of receipt of recent chemotherapy
2. Patients with minimal chance of survival and life expectancy less than 3-5 days as defined by an APACHE II score of ≥ 35 at time of consideration for study eligibility
3. Patients with history or current evidence of autoimmune disease including for example: myasthenia gravis, Guillain Barre syndrome, systemic lupus erythematosus, multiple sclerosis, scleroderma, ulcerative colitis, Crohn's disease, autoimmune hepatitis, Wegener's etc.
4. Patients who have received a solid organ transplant or bone marrow transplant.
5. Patients with active or a history of acute or chronic lymphocytic leukemia
6. AIDS-defining illness (category C) diagnosed within the last 12 months prior to study entry
7. Known history of chronic HBV infection and not on treatment with HBV nucleoside analogues prior to the current hospitalization or HBV DNA > 100 IU/mL
8. Known history of infection with HCV and currently undergoing treatment for HCV infections or has detectable HCV RNA
9. Known history of tuberculosis and currently undergoing treatment for tuberculosis
10. History of splenectomy
11. Any hematologic disease associated with hypersplenism, such as thalassemia, hereditary spherocytosis, Gaucher's Disease, and autoimmune hemolytic anemia
12. Participation in another investigational interventional study testing a drug or a medical device within the last 3 months prior to study entry
13. Patients receiving immunosuppressive drugs, e.g., TNF-alpha inhibitors, for any reason, or systemic corticosteroids other than hydrocortisone at a dose of 300 mg/day
14. Patients receiving concurrent immunotherapy or biologic agents; including growth factors, cytokines and interleukins other than the study medication : IL-2, Interferons α, β and γ, GM-CSF, G-CSF, HIV vaccines, immunosuppressive drugs, hydroxyurea, immunoglobulins, adoptive cell therapy
15. Prior exposure to IL 7 or other drugs specifically targeting T cells
16. Presence of an advanced directive to withhold or withdraw life-sustaining treatment, DNR order or no CPR order, or comfort measures only order
17. Patients for whom prognosis is poor and source control of septic event is considered unlikely per the clinical and research teams.
18. Patients under guardianship

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Lymphocyte reconstitution | day 29 versus baseline
  Change in absolute lymphocyte count (ALC) of ≥ 50%. If this 50% increase over baseline is reached in the placebo group due to natural immune reconstitution, then the day 29 percent increase of ALC over baseline will be compared between the two groups.

SECONDARY OUTCOMES:
adverse events | 90 days after study treatment initiation
  Incidence and scoring of all grade 3-4 adverse events
Secondary Infections | within 90 days after treatment initiation
  Incidence of secondary infections based on pre-specified criteria as adjudicated by the Secondary Infections Committee (SIC)
Days in the ICU | within 90 days after treatment initiation
  Number of days in ICU following study treatment initiation during the index hospitalization
readmissions to the ICU | within 90 days after treatment initiation
  Number of readmissions to ICU following study treatment initiation during index hospitalization
organ support free days | within 90 days after treatment initiation
  Number of organ support free days (OSFDs) following study treatment initiation during the index hospitalization
re-hospitalization | within 90 days following study treatment initiation
  the incidence of re-hospitalization
Mortality rate | 90 days after study treatment initiation
  All-cause mortality
T cell reconstitution | through day 90
  Absolute numbers of CD4+ and CD8+T-cell counts
Percentage of patients reaching normal ALC | through day 90
  Percentage of patients reaching absolute lymphocyte counts (ALC) > 1200
Quantification of IL-7 receptor | through day 90
  Effects on soluble and cellular IL-7 receptor (CD127) expression
Quantification of HLA-DR on monocytes | through day 90
  Effects on circulating monocyte HLA-DR expression
Change of IL-6 blood levels | through day 90
  Effects on whole blood circulating cytokines IL-6
Change of IL-10 blood levels | through day 90
  Effects on whole blood circulating IL-10
Change of TNF-α blood levels | through day 90
  Effects on whole blood circulating TNF-α
CYT107 Pharmacokinetic Tmax | Day 1 and Day 15
  determination of Tmax
CYT107 Pharmacokinetic Cmax | Day 1 and Day 15
  determination of Cmax
CYT107 Pharmacokinetic half life | Day 1 and Day 15
  determination of half-life
CYT107 Pharmacokinetic clearance | Day 1 and Day 15
  determination of clearance
CYT107 Pharmacokinetic area under curve | Day 1 and Day 15
  determination of area under curve
anti-CYT107 antibodies | day 1, day 29 or hospital discharge, day 90 and day 180 if previous sample positive
  Quantification of circulating anti-CYT107 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hotchkiss, MD, Principal Investigator — Washington University School of Medicine; Bruno François, MD, Principal Investigator — Limoges Hospital
Locations (10):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Washington University School of Medicine, St Louis, Missouri
- France (8):
  - CHU Angers, Angers
  - Hopital HENRI MONDOR, Créteil
  - CHU Dijon Bourgogne, Dijon
  - University Hospital of Limoges, Limoges
  - Hôpital Edouard Herriot, Lyon
  - Chr Orleans, Orléans
  - Hopital COCHIN, Paris
  - Chru Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No
Study results will be published Individual data can't be shared and are protected by the new GDPR rule

REFERENCES:
- [Background] Francois B, Jeannet R, Daix T, Walton AH, Shotwell MS, Unsinger J, Monneret G, Rimmele T, Blood T, Morre M, Gregoire A, Mayo GA, Blood J, Durum SK, Sherwood ER, Hotchkiss RS. Interleukin-7 restores lymphocytes in septic shock: the IRIS-7 randomized clinical trial. JCI Insight. 2018 Mar 8;3(5):e98960. doi: 10.1172/jci.insight.98960. PMID 29515037
- [Derived] Daix T, Mathonnet A, Brakenridge S, Dequin PF, Mira JP, Berbille F, Morre M, Jeannet R, Blood T, Unsinger J, Blood J, Walton A, Moldawer LL, Hotchkiss R, Francois B. Intravenously administered interleukin-7 to reverse lymphopenia in patients with septic shock: a double-blind, randomized, placebo-controlled trial. Ann Intensive Care. 2023 Mar 12;13(1):17. doi: 10.1186/s13613-023-01109-w. PMID 36906875